CLINICAL TRIAL: NCT03216967
Title: Multicenter Randomized Two-arms Study Evaluating the BK Viral Clearance in Kidney Transplant Recipients With BK Viremia After Reduction of Immunosuppression Alone vs. Reduction of Immunosuppression and Replacement of Mycophenolate Mofetil by Everolimus
Brief Title: Multicenter Randomized Two-arms Study Evaluating the BK Viral Clearance in Kidney Transplant Recipients With BK Viremia.
Acronym: BK EVER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6646
Record Dates: First submitted 2017-07-04; First posted 2017-07-13 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: BK Virus Nephropathy After Kidney Transplantation
MeSH Terms: interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IS lowering alone (Active Comparator): 50% decrease of the dose of mycophenolic acid at M1 (target AUC 20 mg.h/L)
  Interventions: Drug: everolimus
- Everolimus + IS lowering (Experimental): Stop mycophenolate acid (Cellcept or myfortic) Introduction of everolimus : 2 x 0.75 mg/d per os in patiens treated by ciclosporine
  Interventions: Drug: everolimus

INTERVENTIONS:
Drug: everolimus — Patients with viremia above 2.8 log of copies/ml will be randomized (ratio 1:1) into either of 2 groups Group 1 : control group : immunosuppression lowering or Group 2 : experimental group : immunosuppression lowering and replacement of mycophenolate acid by everolimus Evolution of BKV viremia and allograft function will be assessed during 2 years after randomization

SUMMARY:
BK virus nephropathy (BKVN), a consequence of the strong immunosuppressive therapy given after kidney transplantation, represents a growing problem in the kidney transplant (KT) setting. In recent cohorts, BKVN concerns up to 10% of kidney transplant recipients and early signs of BK virus (BKV) infection as development of asymptomatic viruria and viremia are even much more frequent (40% and 20% of patients, respectively). In this context, finding strategies to prevent BKV infection or treat patients before the occurrence of BKV nephropathy is challenging. For several years, detection of BKV replication by real-time PCR in urine and/or blood of kidney transplant recipients at early stages of infection allowed adaptation of their therapy. As BKV reactivates essentially in patients with over-immunosuppression, the first step of the treatment is the reduction of immunosuppression. However, reducing immunosuppression (IS) can lead to acute rejection and allograft loss. Other treatments have been proposed (cidofovir, quinolones) but their toxicity profile or their lack of clinical efficacy are now demonstrated. Hence, an efficient and safe strategy against uncontrolled BKV replication is urgently needed. MTor-inhibitors are well known immunosuppressive drugs used in organ transplantation to prevent graft-rejection. They have furthermore anti-viral effects that can be beneficial for prevention of viral infections after transplantation. Recent evidence that inhibition of mTor pathway had an impact on BK infected cells provides additional insight into the observed benefits associated with these drugs. The aim of our study is to evaluate the effect of the mTor inhibitor everolimus on the prevention of severe BKV infection (BKV nephropathy or loss of the allograft) after kidney transplantation compared to the reduction of immunosuppression alone in kidney recipients with BK viremia.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Kidney transplant recipients
* Patients treated by a calcineurin inhibitor and mycophenolic acid
* Viremia >= 2.8 log UI/ml
* Patients who have given written informed consent
* Negative pregnancy test (blood β-HCG dosage)

Exclusion Criteria:

* Known proved BKV nephropathy
* Hypersensitivity to everolimus, sirolimus or excipient
* Concomitant treatment by leflunomide, cidofovir, sirolimus, Millepertuis (Hypericum Perforatum)
* Pregnant or lactating women
* Women of child bearing potential unless they are using a birth control method

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
The main objective of our study is to evaluate the proportion of patients with BKV clearance 6 months after introduction of everolimus in kidney recipients who develop BKV viremia compared to patients managed with IS reduction alone | 6 months after randomization
  The primary end point is the proportion of patients with clearance of BK viremia assessed by blood PCR and functional graft 6 months after modification of immunosuppressive therapy

CONTACTS AND LOCATIONS:
Locations (15):
- France (15):
  - CHU - Hôpital Sud, Amiens
  - CHRU d'Angers, Angers
  - CHU - Hôpital de la Cavale Blanche, Bois-Guillaume
  - CHU - Hôpital de la Cavale Blanche, Brest
  - CHU Côte de Nacre, Caen
  - CHU Hôpital Gabriel Montpied, Clermont-Ferrand
  - CHU - Hôpital Dupuytren, Limoges
  - Hôpital Edouard Herriot, Lyon
  - AP-HP Hôpital Necker, Paris
  - AP-HP - Hôpital Georges Pompidou, Paris
  - CHU Poitiers - Hôpital Jean Bernard, Poitiers
  - CHU - Hôpital Maison Blanche, Reims
  - CHU Rennes - Hôpital Pontchaillou, Rennes
  - Les Hôpitaux Universitaires, Strasbourg
  - CHRU - Hôpital Bretonneau, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Caillard S, Meyer N, Solis M, Bertrand D, Jaureguy M, Anglicheau D, Ecotiere L, Buchler M, Bouvier N, Schvartz B, Rerolle JP, Heng AE, Couzi L, Duveau A, Morelon E, LeMeur Y, Golbin L, Thervet E, Benotmane I, Fafi-Kremer S. Insights from the BKEVER Trial comparing everolimus versus mycophenolate mofetil for BK Polyomavirus infection in kidney transplant recipients. Kidney Int. 2025 Feb;107(2):338-347. doi: 10.1016/j.kint.2024.09.018. Epub 2024 Oct 28. PMID 39490986